CLINICAL TRIAL: NCT04045106
Title: The Acute Effect of Proprioceptive Neuromuscular Facilitation on Cervical Range of Motion, Strength and Proprioception
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 10269393
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Proprioception; Neck
Keywords: Proprioception; Proprioceptive Neuromuscular Facilitation,; Cervical spine; stretching
MeSH Terms: interventions — Muscle Stretching Exercises; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNF pattern (Experimental): PNF patterns were performed using Dynamic of reversals technique which is characterized as active motion alternating from one direction (agonist) to the opposite (antagonist) without relaxing. The cervical patterns consisted of
  1. Cervical flexion with right rotation followed by extension with left rotation.
  2. Cervical flexion with left rotation followed by extension with right rotation.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Patterns
- PNF stretching (Experimental): PNF stretching was done using contract-relax-antagonist contract (CRAC) technique for cervical flexors, extensors, right and left lateral flexors, right rotators and left rotators.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation stretching
- control (Sham Comparator): Participants allocated to the control group received ineffective passive ROM.
  Interventions: Other: Passive range of motion

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation Patterns — The participants were asked to sit on a chair, the therapist performed the pattern of movement himself then passively applied the pattern on the participant then asked the participant to perform the pattern, and the therapist observed and corrected the movement if it was done improperly.Then participants were told that the therapist will resist their movement, they were also told to keep breathing normally and to report any discomfort and/or pain.After mastering the pattern,the therapist placed one hand on the participant's mandibular and the other hand approximately between parietal and occipital bones to apply resistance through out the ROM, each pattern performed for 3 sets of 10 repetitions with 1-2-minute rest between sets.
  Arms: PNF pattern
Other: Proprioceptive Neuromuscular Facilitation stretching — was done for 6 repetitions with hold for 6 seconds in position of stretch and sub maximal isometric contraction for 6 seconds, 1-2-minute rest was given before changing the target muscle group
  Arms: PNF stretching
Other: Passive range of motion — ineffective passive ROM for 10 repetitions for flexion, extension, right and left side bending and right and left rotation, it was done from neutral position to the limit of motion without causing any stretch to the muscle.
  Arms: control

SUMMARY:
the aim of the study was to investigate the immediate influence of proprioceptive neuromuscular facilitation on cervical range of motion, strength and proprioception

DETAILED DESCRIPTION:
the study evaluates the influence of two proprioceptive neuromuscular facilitation techniques (PNF patterns and PNF stretching) on cervical proprioception. PNF techniques are regularly used techniques among physiotherapist. also there is a lack of studies that investigated the effect of PNF on cervical proprioception

ELIGIBILITY:
Inclusion Criteria:

* Neck disability index score of 5 or less
* Able to understand and follow instructions
* Above 18 years old

Exclusion Criteria:

* Cervical trauma
* History of cervical inter-vertebral disc pathology
* Rheumatic diseases
* Whiplash syndrome
* History of surgeries to the neck, face and shoulders
* History of systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Cervical Proprioception: Joint position accuracy method using cervical range of motion instrument. | 1 day
  Joint position accuracy method using cervical range of motion instrument. Participants were asked to sit and put on the CROM instrument, then they were instructed to start moving their head to one of directions then the assessor stopped them at 30 degrees and told them to feel the amount of movement and muscle tension, this was repeated 3 times as a reference, then they were asked to do the movement with the eyes closed until they reach the target angle, this was repeated for 3 times, this was done for each direction and the assessor recorded the results. Cervical proprioception was done for flexion, extension, right side bending, left side bending, right and left rotation

SECONDARY OUTCOMES:
Range Of Motion | 1 day
  Active Range of motion (AROM) was measured using cervical range of motion instrument.
  CROM instrument were placed on the participants head, then the assessor asked the participant to move towards the movement direction until they reach the limit.
Muscle strength | 1 day
  The measurement were taken for cervical flexors, extensors, right and left rotators, right and left side benders, each was done in an against gravity position.

CONTACTS AND LOCATIONS:
Overall Officials: SULE DEMIRBASISTANBUL, Study Director — Yeditepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Yeditepe University, Ataşehir, Istanbul
  - Bahcesehir University, Beşiktaş, Istanbul

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04045106/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04045106/ICF_001.pdf